CLINICAL TRIAL: NCT04597346
Title: A Single-arm, Prospective, Multicenter, Real-world Study to Evaluate the Safety and Efficacy of Bronchoscopic Transparenchymal Nodule Access (BTPNA) for the Diagnosis of Peripheral Lung Lesions
Brief Title: Evaluate the Diagnostic Value of BTPNA for PPL: a Real-world Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Henan Provincial People's Hospital (Other); Beijing Chao Yang Hospital (Other); Shandong Public Health Clinical Center (Other Government); West China Hospital (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Xi 'an International Medical Center Hospital (Unknown); Emergency General Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital
Other Study IDs: SHCHE202003
Record Dates: First submitted 2020-10-14; First posted 2020-10-22 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Peripheral Pulmonary Lesion
Keywords: Bronchoscopic Transparenchymal Nodule Access; Peripheral Pulmonary Lesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Bronchoscopic Transparenchymal Nodule Access — Bronchoscopic Transparenchymal Nodule Access (BTPNA) is locating the lesion in the lung tissue guided by the bronchoscope navigation system (LungPro) in the natural lumen (bronchus), and automatically calculates the best point of entry (POE) and the best route to avoid blood vessels. An opening is made from the POE under the endoscope, and is extended with a balloon dilator. Combined with X-ray fluoroscopy, a sheath with a blunt-tip core is used in the lung parenchyma to reach the lesion site, and then biopsy diagnosis or treatment.

SUMMARY:
The study is designed as a multicenter prospective trial of BTPNA for the diagnosis of peripheral pulmonary lesions in the real world. The purpose of the study is to evaluate the safety and effectiveness of BTPNA and to explore the factors of diagnosis rate.

DETAILED DESCRIPTION:
The study will be conducted at about 10 clinical centers. Patients will be first screened, and only after meeting all the selection criteria, not meeting any exclusion criteria, and signing the informed consent, could they be enrolled in the group to receive BTPNA to sample the target lesions. The primary endpoint is the diagnostic yield of BTPNA. The secondary endpoints include the success rate of navigation, the operation time of the bronchoscope and so on.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years old.
2. Newly diagnosed patients whose chest CT shows peripheral pulmonary lesions that have bronchus signs but are difficult to reach through the intrabronchial path, or are adjacent to the airway, or have no bronchus sign, and are suspected of malignancy which need non-surgical biopsies.
3. The diameter of the lesions is greater than or equal to 0.8cm and less than 5cm
4. The location of lesions results in the following situations where transthoracic needle aspiration (TTNA) is difficult to obtain a diagnosis or the operation is relatively risky, or have not been diagnosed by TTNA and other non-surgical biopsies in the past.
5. Lesions can be accessed by BTPNA technology in preoperative assessment.
6. Understand the research and sign the informed consent form.

Exclusion Criteria:

1. Contraindications for bronchoscopy.
2. The lesions are adjacent to the target trachea or bronchus of points of entry(POE).
3. Severe cardiopulmonary dysfunction and other diseases that may significantly increase the risk of surgery.
4. Routine bronchoscopy showed visible lesions in the lumen.
5. The investigator believes that the patient has other conditions that are not suitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed patients whose chest CT showed suspect malignant peripheral lung lesion and are scheduled to receive non-surgical biopsies with lesion access via BTPNA.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | Six months
  Diagnostic yield is defined as the proportion of lesions diagnosed by BTPNA in all lesions undergoing bronchoscopy biopsy by BTPNA.

SECONDARY OUTCOMES:
The success rate of navigation | Immediately after bronchoscopic biopsy
  The success rate of navigation is defined as the proportion of the number of lesions confirmed by ultrasound (and/or fluoroscopy) to the number of lesions in all BTPNA guided by the navigation system.
The success rate of biopsy | Immediately after bronchoscopic biopsy
  The success rate of biopsy is the number of lesions obtained by using BTPNA biopsy to obtain at least one qualified abnormal lung tissue sample that can be used for pathological diagnosis, divided by the total number of lesions obtained using BTPNA biopsy.
The operation time of the bronchoscope | Immediately after bronchoscopic biopsy
  The operation time of the bronchoscope is defined as the total time from insertion of the bronchoscope to withdrawal of the bronchoscope, not including the operation time of EBUS-TBNA.
The total time of lesion access | Immediately after bronchoscopic biopsy
  The total time of lesion access is defined as the total time from the insertion of the bronchoscope to the arrival confirmed by ultrasound probes (and/or fluoroscopy).
The intraoperative fluoroscopy time | Immediately after bronchoscopic biopsy
  The intraoperative fluoroscopy time is defined as the total fluoroscopy time (fluoroscopy reading) between the insertion of the bronchoscope and the withdrawal of the bronchoscope.
Factors affecting the diagnosis rate | Six months
  Factors affecting the diagnosis rate, including the size of the lesions, the bronchial signs, the location of the lesions and so on will be analyzed.
Factors affecting the biopsy success rate | Six months
  Factors affecting the biopsy success rate, including the size of the lesions, the bronchial signs, the location of the lesions and so on will be analyzed.
Factors affecting the navigation success rate | Six months
  Factors affecting the navigation success rate, including the size of the lesions, the bronchial signs, the location of the lesions and so on will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD, PhD, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chechani V. Bronchoscopic diagnosis of solitary pulmonary nodules and lung masses in the absence of endobronchial abnormality. Chest. 1996 Mar;109(3):620-5. doi: 10.1378/chest.109.3.620. PMID 8617067
- [Result] Baaklini WA, Reinoso MA, Gorin AB, Sharafkaneh A, Manian P. Diagnostic yield of fiberoptic bronchoscopy in evaluating solitary pulmonary nodules. Chest. 2000 Apr;117(4):1049-54. doi: 10.1378/chest.117.4.1049. PMID 10767238
- [Result] Tamiya M, Okamoto N, Sasada S, Shiroyama T, Morishita N, Suzuki H, Yoshida E, Hirashima T, Kawahara K, Kawase I. Diagnostic yield of combined bronchoscopy and endobronchial ultrasonography, under LungPoint guidance for small peripheral pulmonary lesions. Respirology. 2013 Jul;18(5):834-9. doi: 10.1111/resp.12095. PMID 23586738
- [Result] Gilbert C, Akulian J, Amador RO, Lee H, Yarmus L. Novel bronchoscopic strategies for the diagnosis of peripheral lung lesions: present techniques and future directions. Respirology. 2014 Jul;19(5):636-44. doi: 10.1111/resp.12301. Epub 2014 May 6. PMID 24797257
- [Result] Sterman DH, Keast T, Rai L, Gibbs J, Wibowo H, Draper J, Herth FJ, Silvestri GA. High yield of bronchoscopic transparenchymal nodule access real-time image-guided sampling in a novel model of small pulmonary nodules in canines. Chest. 2015 Mar;147(3):700-707. doi: 10.1378/chest.14-0724. PMID 25275338
- [Result] Herth FJ, Eberhardt R, Sterman D, Silvestri GA, Hoffmann H, Shah PL. Bronchoscopic transparenchymal nodule access (BTPNA): first in human trial of a novel procedure for sampling solitary pulmonary nodules. Thorax. 2015 Apr;70(4):326-32. doi: 10.1136/thoraxjnl-2014-206211. Epub 2015 Mar 6. PMID 25746631
- [Result] Harzheim D, Sterman D, Shah PL, Eberhardt R, Herth FJ. Bronchoscopic Transparenchymal Nodule Access: Feasibility and Safety in an Endoscopic Unit. Respiration. 2016;91(4):302-6. doi: 10.1159/000445032. Epub 2016 Mar 24. PMID 27007334